CLINICAL TRIAL: NCT04827953
Title: Phase Ib/IIa Study to Evaluate Safety and Efficacy of Treatment With the Hedgehog Inhibitor NLM-001 and Chemotherapy (Gemcitabine and Nab-Paclitaxel) Plus Zalifrelimab as First Line Treatment in Patients With Advanced Pancreatic Cancer
Brief Title: Study to Evaluate the Safety and Efficacy of Treatment With NLM-001 and Standard Chemotherapy Plus Zalifrelimab in Patients With Advanced Pancreatic Cancer
Acronym: NUMANTIA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nelum Corp (Industry)
Collaborators: Apices Soluciones S.L. (Industry); Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLM-2020-01 / NUMANTIA; 2020-004932-52 (EudraCT Number)
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational treatment (Experimental): Conventional Chemotherapy (Gemcitabine + nab-paclitaxel) plus NLM-001 plus Zalifrelimab
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel; Drug: NLM-001; Drug: Zalifrelimab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV on days 1, 8 and 15 (conventional chemotherapy).
Drug: Nab paclitaxel — Nab-Paclitaxel 125 mg/m2 IV on days 1, 8 and 15 (conventional chemotherapy).
Drug: NLM-001 — NLM-001 will be administered three cycles consecutively followed by two rest cycles.
Drug: Zalifrelimab — Zalifrelimab administration each 6 weeks.

SUMMARY:
In order to improve the survival rates and decrease progression of pancreatic advanced cancer, this study aims to evaluate the first line treatment approved for this disease (gemcitabine plus nab-paclitaxel) in combination with two experimental drugs, an inhibitor of the signaling pathway of Hedgehog and an immunotherapy drug able of blocking the CTLA-4 receptor.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the leading neoplasms in the world in terms of mortality, with very low survival rates mainly due to its rapid progression and diagnosis in advanced stages, which makes its treatment extremely difficult.

Gemcitabine plus nab-paclitaxel is currently considered the first-line standard treatment for advanced pancreatic cancer due to this superiority against other treatments.

In order to find an alternative to improve survival of advanced pancreatic cancer, this study aims to evaluate the efficacy with first-line treatment in combination of two experimental drugs, a Hedgehog pathway inhibitor (NLM-001) and a CTLA-4 blocker (zalifrelimab) in previously untreated patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Investigators must ensure that patients are able to understand the requirements of the study and provide informed consent
2. Age ≥18 years
3. Histological or cytological diagnosis of pancreatic adenocarcinoma
4. Stage IV disease
5. No prior treatment for advanced disease. Patients who have received chemotherapy for localize disease are eligible if at least six months have elapsed from the last chemotherapy treatment
6. Measurable disease per RECIST 1.1 as determined by the investigator
7. ECOG (Eastern Cooperative Oncology Group) PS 0-1
8. Sufficient hematopoietic, renal and liver function as defined as:

   * Neutrophil count ≥ 1.5 x 10*9 / L
   * Platelet count ≥ 100 x 10*9 / L
   * Bilirubin ≤ 1.5 x ULN (upper limit of normal)
   * AST and / or ALT ≤2.5 x ULN or ≤5 for patients with liver disease
   * Serum creatinine ≤ 1.5 x ULN
9. Tumor lesion amenable for safe repeated biopsy
10. Women of child-bearing age and men who wish to participate in the study must agree to use appropriate contraceptive methods from the signing of informed consent until 3 months after discontinuation of the study drug

    * Adequate contraception includes abstinence, oral contraceptives, transdermal patches, and injections that prolong release of a progestogen (starting at least 4 weeks prior to the administration of the investigational drug), double barrier method: condom or female condom (diaphragm or condom / vaginal) plus spermicide, intrauterine device (IUD), implant or a vaginal ring (placed at least 4 weeks prior to administration of investigational drug) or male partner sterilization (vasectomy with documentation of azoospermia) before the inclusion of the woman in the trial if the male is the only sex partner of the woman

Investigators must ensure that patients recruited will be able to meet all study requirements, including tumor biopsy, chemotherapy and monitoring

Exclusion Criteria:

1. Active or uncontrolled infection, disease or serious medical condition that may interfere with the patient's eligibility or treatment
2. History of psychiatric condition that would compromise the patient's ability to understand or comply with the requirements of the protocol, or the ability to provide informed consent
3. Concurrent antineoplastic therapy
4. Pregnant or lactating women
5. History of allergic reactions attributed to compounds of similar chemical structure or similar biological study drug composition
6. History of life-threatening serious adverse events to Gemcitabine or Nab-Paclitaxel
7. Prior chemotherapy or chemo-radiation therapy for advanced pancreatic cancer
8. Patients requiring or being treated with potent CYP3A4 inhibitors and inducers
9. Other malignancies treated within the last 5 years, except in situ cervix carcinoma or nonmelanoma skin cancer
10. History of interstitial lung disease
11. Subjects with a history or presence of a known clotting disorder or difficulty achieving haemostasis will be excluded
12. Primary or secondary immunodeficiency, including immunosuppressive disease or autoimmune disease (including autoimmune endocrinopathies).

    Note: Subjects with diabetes type 1, vitiligo, psoriasis, hypo-, or hyperthyroid disease not requiring immunosuppressive treatment are eligible. Subjects with Type 2 diabetes mellitus are allowed
13. Subjects with a known history of human immunodeficiency virus 1 and 2, human T lymphotropic virus 1.
14. Administration of anticancer medications or investigational drugs within the following intervals before the first administration of study drug:

    1. A 1-week washout is permitted for palliative radiation to non- central nervous system (CNS) disease, with medical monitor approval. Subjects must also not have had radiation pneumonitis as a result of treatment and cannot participate in the study if they are on chronic corticosteroids for radiation pneumonitis Note: Bisphosphonates and denosumab are permitted medications
    2. ≤7 days for prior corticosteroid treatment, with the following exceptions:

       * Use of an inhaled or topical corticosteroid is permitted
       * Corticosteroid premedication for radiographic imaging for dye allergies is permitted
       * Use of physiologic corticosteroid replacement therapy may be approved after consultation with the medical monitor
    3. ≤7 days for immunosuppressive-based treatment for any reason, with the exceptions noted above for prior corticosteroid treatment
    4. ≤21 days or 5 half-lives before first dose of study treatment for all other investigational study drugs or devices. For investigational agents with long half-lives (e.g., >5 days), enrollment before the fifth half-life requires medical monitor approval
15. Has not recovered to grade ≤1 from toxic effects of prior therapy and/or complications from prior surgical intervention before starting therapy Note: Subjects with grade ≤2 neuropathy and alopecia are an exception and may enroll
16. History or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful
17. Concurrent participation in other investigational drug trials
18. Known central nervous system (CNS) involvement as follows:

    * Untreated CNS metastases.
    * Leptomeningeal metastases. Note: Patients may be eligible if CNS metastases have been treated and patients have neurologically returned to baseline (except for residual signs and symptoms related to the CNS treatment).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy according to response | 17 months
  Objective Response Rate (ORR): Complete Response (CR) + Partial Response (PR) according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Frequency of occurrence of adverse events | 8 months
  Frequency of occurrence of adverse events according to NCI-CTCAE v5.0 criteria
Treatment efficacy according to disease control rate | 8 months
  Disease Control Rate (DCR): Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) evaluated by RECIST 1.1 criteria
Treatment efficacy according to progression free survival (PFS) | 8 months
  Time in months from the patient's study enrolment until patient progression according to RECIST 1.1 criteria or death.
Treatment efficacy according to Duration of Response (DoR) | 8 months
  Time between the date of first confirmed response to the date of the first documented tumor progression (per RECIST 1.1), or death due to any cause, whichever occurs first
Treatment efficacy according to Overall Survival (OS) | 8 months
  Time in months since the patient's study enrolment until death.
CA 19.9 | 8 months
  Decrease in CA 19.9 levels > 50%
Gli mRNA and SMA + CAF expression and ORR | 1 month
  Correlation between change in Gli mRNA and SMA + CAF expression and Objective Response Rate (ORR).
Gli mRNA and SMA + CAF expression and PFS | 1 month
  Correlation between change in Gli mRNA and SMA + CAF expression and Progression Free Survival (PFS).
Collagen structure and ORR | 1 month
  Correlation between change in Collagen structure and Objective Response Rate (ORR)
Collagen structure and PFS | 1 month
  Correlation between change in Collagen structure and Progression Free Survival (PFS).
Lymphocyte infiltration and ORR | 1 month
  Correlation between change in lymphocyte infiltration and Objective Response Rate (ORR).
Lymphocyte infiltration and PFS | 1 month
  Correlation between change in lymphocyte infiltration and Progression Free Survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Macarulla, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (6):
- Spain (6):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Virgen De La Victoria, Málaga, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitario Marqués del Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: No